CLINICAL TRIAL: NCT06927817
Title: The Effect of Hyoscine-N-Butylbromide on Nausea and Pain in Laparoscopic Cholecystectomy: A Prospective Randomized Study
Brief Title: The Effect of Hyoscine-n-butylbromide on Nausea and Pain in Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Süheyla Abitağaoğlu, Associate Professor, MD, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: no sponsorship
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Cholecystitis; Pain; Nausea
Keywords: Hyoscine N-Butylbromide; Laparoscopic Cholecystectomy; Ondansetron; Pain; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Cholecystitis; Pain; Nausea; Postoperative Nausea and Vomiting | interventions — Butylscopolammonium Bromide; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hyoscine-n-butylbromide (Experimental): after removal of gall bladder 20mg hyoscine-n-butylbromide in 100ml saline wİll be administered
  Interventions: Drug: hyoscine-n-butylbromide, ondansetron
- ondansetron (Active Comparator): 4mg ondansetron infusion in 100ml saline was administered
  Interventions: Drug: • hyoscine-n-butylbromide • ondansetron

INTERVENTIONS:
Drug: hyoscine-n-butylbromide, ondansetron — In patients in Group Hyoscine 20mg hyoscine-n-butylbromide in 100ml saline and in Group Ondansetron 4mg ondansetron infusion in 100ml saline will be administered in Group-O. The patients will be followed-up in terms of nausea, vomiting, and pain at the postoperative 15th, and 30th minutes and at the 3rd, 6th, 12th, and 24th hours.
  Other Names: • hyoscine-n-butylbromide • ondansetron
  Arms: hyoscine-n-butylbromide
Drug: • hyoscine-n-butylbromide • ondansetron — In patients in Group Hyoscine 20mg hyoscine-n-butylbromide in 100ml saline and in Group Ondansetron 4mg ondansetron infusion in 100ml saline will be administered in Group-O. The patients will be followed-up in terms of nausea, vomiting, and pain at the postoperative 15th, and 30th minutes and at the 3rd, 6th, 12th, and 24th hours.
  Arms: ondansetron

SUMMARY:
The goal of this randomized double blind study is to compare the effects of hyoscine-n-butylbromide, and ondansetron on postoperative nausea-vomiting, and pain in patients who underwent laparoscopic cholecystectomy.The main questions it aims to answer are:

1. Is antiemetic properties of hyoscine-n-butylbromide effective after laparoscopic cholecyctectomy?

1. Does hyoscine-n-butylbromide have valuable effects on postoperative pain after laparoscopic cholecyctectomy?

Participants will be the paients undergoing laparoscopic cholecyctectomy.

The patients participating in the study were randomized into two groups as Group-HBB, and Group-O.

After the gallbladder removed, IV infusion of 1000 mg paracetamol, and 1.5 mg/kg tramadol will administered to the patients. 20 mg hyoscine-n-butylbromide in 100 ml saline will administered to the patients in Group-HBB, and 4 mg ondansetron infusion in 100 ml saline will be administered to the patients in Group-O.

Postoperative nausea and vomitting score and pain intensity and rescue drugs will be recorded in postoperative 24 hours.

DETAILED DESCRIPTION:
After obtaining the informed consent form from the patients, a total of 134 patients undergoingt laparoscopic cholecystectomy surgery will be inclueded in the study. The patients participating in the study will be randomized into two groups as Group-HBB, and Group-O by the closed envelope method. The patients will be blinded to groups they belonged to. Routine peripheral oxygen saturation, noninvasive blood pressure, electrocardiography, and bispectral index (BIS) monitoring will be performed.. BIS-guided 2-2.5mg/kg propofol, and 2mcg/kg fentanyl intravenously, and 0.6mg/kg rocuronium injection will be administered. In order to maintain the BIS value between 40-60, 1-2% sevoflurane inhalation in 40/60% oxygen/air mixture in 2-liter flow, and 0.1-0.5mc/kg/min remifentanil infusion will be applied. After the gallbladder removed, IV infusion of 1000 mg paracetamol, and 1.5 mg/kg tramadol will administered to the patients. 20 mg hyoscine-n-butylbromide in 100 ml saline will administered to the patients in Group-HBB, and 4 mg ondansetron infusion in 100 ml saline will be administered to the patients in Group-O. After the surgery terminates, 2 mg/kg sugammadex will be used to antagonize the muscle relaxant effect, and patients with adequate respiratory effort, and a BIS value above 85 will be extubated.

Demographic data of the patients such as age, body mass index, gender, comorbidities, ASA score, and smoking status will be recorded. Nausea, vomiting, and pain status will be examined in the recovery unit at postoperative 15th, and 30th minutes and in the ward at the 3rd, 6th, 12th and 24th hours. Follow-ups will be performed by an anesthesiologist who is blind to groups of the patients. A 4-point scale will be used for nausea-vomiting (0: no nausea and vomiting, 1: nausea, no vomiting, 2: nausea, vomiting, 3: vomiting more than twice), and a 10 cm VAS score will be used for assessig the pain level. Patients with a pain level of 4 and above will be administered 20 mg of tenoxicam intravenously as an analgesic. If the nausea score is >0, 10 mg metoclopramide iv will be administered, and if the score was still >0 after 30 minutes, 4 mg dexamethasone iv will be administered.

ELIGIBILITY:
Inclusion Criteria:

ASA score of 1-2 who undergoing laparoscopic cholecystectomy 18-65 years of age

Exclusion Criteria:

* Patients who are allergic to the drugs used in the study, have an ASA score of 3-4, congestive heart failure or arrhythmia, motion sickness, central nervous system pathology, glaucoma, prostate hypertrophy, and a body mass index above 35, and used antihistamines will not included in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
postoperative nausea and vomiting | 15th, and 30th minutes and at the 3rd, 6th, 12th, and 24th hours.
  A 4-point scale will be used for nausea-vomiting (0: no nausea and vomiting, 1: nausea, no vomiting, 2: nausea, vomiting, 3: vomiting more than twice)
Postoperative pain | 15th, and 30th minutes and at the 3rd, 6th, 12th, and 24th hours.
  10 cm VAS score will be used for assessig the pain level

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Fatih Sultan Mehmet Health Research and Application Center,, Istanbul, Istanbul, Turkey (Türkiye)